CLINICAL TRIAL: NCT02238366
Title: A Non-interventional, Multi-centric, Observational, Prospective Study to Collect the Criteria on Which Renewal of GnRH Analogue Treatment With Triptorelin (Diphereline 3.75mg or Diphereline pr 11.25mg) is Made in Patients Recently Diagnosed With Prostate Cancer Requiring Androgen Deprivation Therapy
Brief Title: Study To Assess Renewal Of Treatment In Patients Recently Diagnosed With Prostate Cancer
Acronym: CHRONOS3
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-52014-213
Record Dates: First submitted 2014-09-02; First posted 2014-09-12 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate; Injections, Intramuscular; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prostate cancer patients: Patients recently diagnosed with prostate cancer requiring ADT.
  Interventions: Drug: triptorelin

INTERVENTIONS:
Drug: triptorelin — This is an observational study. Thus, the treatment selection with triptorelin (Diphereline® or Diphereline PR®) is at investigator's discretion based on the current practice principles and guidelines/protocols, in accordance with the Summary of Product Characteristics (SmPC) approved in Romania by the National Medicines Agency.
  Other Names: Diphereline 3.75mg or Diphereline PR (prolonged release) 11.25mg intramuscular (IM.) Injection

SUMMARY:
The purpose of this study is to collect some parameters which may help to provide guidance on how Androgen Deprivation Therapy (ADT) drugs are renewed and physician satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult men, ≥18 years old, with recently diagnosed locally advanced or metastatic prostate cancer scheduled to receive androgen deprivation therapy as monotherapy or as concomitant and adjuvant therapy in association with radiation therapy, with a 1 or 3 month GnRH analogue triptorelin formulation
* Expected survival > 12 months.
* Patients having provided written informed consent.
* Patients mentally fit for completing a questionnaire.

Exclusion Criteria:

* Treatment with any investigational drug within the last 3 months before study entry or planning to participate in a study.
* Patients who already have been treated with a GnRH analogue within the last year.
* Patients with hypersensitivity to GnRH, GnRH analogue, triptorelin or its excipients.
* Patients with a contraindication according to SmPC.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men recently diagnosed with locally advanced or metastatic prostate cancer receiving ADT.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2013-11; Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients for whom the initial Gonadotropin-releasing Hormone (GnRH) analogue formulation has been renewed. | 1 month
  To evaluate the percentage of patients for whom the initial GnRH analogue formulation has been renewed at 1-month +/- 7 days for Diphereline 3.75mg.
Percentage of patients for whom the initial GnRH analogue formulation has been renewed. | 3 months
  To evaluate the percentage of patients for whom the initial GnRH analogue formulation has been renewed at at 3-months +/- 10 days for Diphereline PR 11.25mg (Visit 2).

SECONDARY OUTCOMES:
Percentage of patients for whom the initial GnRH analogue formulation has been renewed at each follow up visit | 6 and 12 months
  To evaluate the percentage of patients for whom the initial GnRH formulation (triptorelin-Diphereline®) had been renewed at each follow up visit [Visit 3 (at 6-months +/- 3 weeks), Visit 4 (at 12-months +/- 6 weeks)].
Percentage of patients that switched from a 1-month to a 3-months formulation | 3, 6, 12 months
  To evaluate the percentage of patients having switched from a 1-month to a 3-months formulation at each visit [Visit 2 (at 1 month or 3 months), Visit 3 (at 6 months +/- 3 weeks), Visit 4 (at 12 months +/- 6 weeks)].

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (7):
- Romania (7):
  - Arad
  - Bucharest
  - Cluj-Napoca
  - Constanța
  - Craiova
  - Iași
  - Timișoara